CLINICAL TRIAL: NCT00467610
Title: A Phase 2, Open-Label, Multiple-Dose Study Investigating the Efficacy and Safety of Panhematin in Patients With Low or Intermediate-1 Risk Myelodysplastic Syndrome
Brief Title: Phase 2, Open-Label, Multi-Dose Study of Panhematin in Patients With MDS
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: lack of efficacy.
Sponsor: Rush University Medical Center (Other)
Collaborators: H. Lundbeck A/S (Industry)
Responsible Party: Principal Investigator, Jamile Shammo, Associate Professor of Medicine and Pathology, Rush University Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MDS 2005-01; 06011001 (Other Grant/Funding Number: Ovation pharmaceuticals)
Record Dates: First submitted 2007-04-26; First posted 2007-04-30 (Estimated); Results first posted 2014-10-24 (Estimated); Last update posted 2014-10-24 (Estimated); Status verified 2014-10

CONDITIONS: Myelodysplastic Syndrome
Keywords: myelodysplastic; MDS; Panhematin; Hemin
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — Hemin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Panhematin (Experimental)
  Interventions: Drug: Panhematin

INTERVENTIONS:
Drug: Panhematin

SUMMARY:
This is a Phase II, open-label clinical trial examining the role of Panhematin® in patients with MDS. The objective of this study is to evaluate the safety and efficacy of Panhematin® (hematin for injection) in the treatment of adult patients (≥ 18 years of age) with low-risk MDS.

The study will be conducted on an outpatient basis and will consist of the following:

* A Screening Period (within 28 days of the Day 1)
* Screening bone marrow aspiration and biopsy up to 60 days prior to receiving study medication
* An 8-week Treatment Period (Days 1 through 4 of Week 1, and weekly visits during Weeks 2 through 8); partial and complete responders in any of the three cell lines may continue treatment for an additional 4 weeks
* A 6-month Post treatment Follow-up Period (monthly clinic visits during Weeks 12 40)

DETAILED DESCRIPTION:
The myelodysplastic syndromes (MDS), a diverse group of hematopoietic stem cell (HSC) disorders, are characterized by ineffective hematopoiesis that manifest clinically as anemia, neutropenia, and/or thrombocytopenia. MDS is most frequently observed in the elderly population (median age between 60 and 70 years) and has a male predominance. The incidence of MDS varies from 2.1 to 12.6 cases per 100,000 people per year, with an estimated prevalence of up to 55,000 patients in the United States [Catenacci, 2005; Williamson, 1994; Aul, 1998; Aul, 2001]. Patients with MDS most frequently present with symptoms of fatigue, pallor, exertional dyspnea, infection, bleeding or bruising [Catenacci, 2005].

MDS can be divided into 2 major subtypes: indolent (or early) MDS, in which pro-apoptotic forces predominate, and aggressive (or advanced) MDS, in which pro-proliferative factors are more common.

The only curative therapy for MDS is allogeneic transplantation [Catenacci, 2005; Thompson, 2005]. Curative treatments are restricted to younger, healthier individuals with histocompatible-matched donors or those able to undergo intensive chemotherapeutic regimens [Catenacci, 2005]. Recently, the FDA approved 3 agents for the treatment of this disease, Vidaza, Dacogen, and revlimid. The latter is approved for a subset of patients with MDS with del 5q abnormality, the former two are more applicable to higher risk disease. Rhu-EPO is currently available to patients with low risk MDS however, if they fail, their options are limited to the agents mentioned above, all of which have significant myelotoxic effects. Effective and less myelosuppressive treatments for low-risk MDS are needed.

We are proposing a novel approach for the treatment of patients with low-risk MDS using heme supplementation with Panhematin® (hemin for injection). Panhematin® is an iron-containing metalloporphyrin, indicated for the amelioration of recurrent attacks of acute intermittent porphyria; it acts to limit the hepatic and/or marrow synthesis of porphyrin, presumably, as a result of the inhibition of aminolevulinic acid synthetase (the enzyme which limits the rate of porphyrin/heme biosynthetic pathway) [Panhematin® Product Prescribing Information].

There are pre-clinical and clinical data to suggest that heme supplementation with Panhematin® (hematin for injection) has potential as a treatment option for patients with MDS. Preliminary data indicate hemin administration has the potential to stimulate progenitor cell growth, stimulate globin synthesis, and elevate overall hemoglobin levels. Panhematin® has been proven to be well tolerated when used therapeutically in patients with acute intermittent porphyria, and it is anticipated to be well tolerated in this patient population. For this study, selected patients will have low or intermediate 1 risk disease by IPSS, and the standard of care for MDS (supportive therapies) will be administered as needed. Measurement of serum porphyrin levels and Hgb F will be done at baseline and at week 8.

ELIGIBILITY:
Inclusion Criteria:

A patient will be eligible for study participation if all of the following criteria are met:

1. The patient must sign and date the IRB/IEC approved Informed Consent Form/HIPAA Authorization prior to study participation.
2. Patient is at least 18 years of age.
3. If female:

   1. Patient, either male or female, is either not of childbearing potential, defined as postmenopausal for at least 1 year or surgically sterile (bilateral tubal ligation, bilateral oophorectomy or hysterectomy), or if of childbearing potential, must comply with an effective method of birth control acceptable to the Investigator during the study (oral contraceptives, Depo-Provera, intra-uterine device), for at least 1 month prior to enrollment and for 1 month following the completion of the study.
   2. Patient is not breastfeeding.
   3. Patient of childbearing potential must have a negative urine or serum pregnancy test during the screening period.
4. Patient has a diagnosis of low- or intermediate-1 risk MDS, as determined by the International Prognostic Scoring (IPSS) (score of 0-1).
5. Patient must be transfusion dependent (i.e., received ≥ 2 units over an 8-week period prior to registration) or have a hemoglobin value ≤ 10 g/dL on the screening laboratories.
6. Patients must have ≤ 10% blasts in the bone marrow and peripheral blood.
7. Patient must have a platelet counts > 50,000/microliters and absolute neutrophil counts (ANC) >500/microliters.
8. Patient must have adequate hepatic and renal functions, defined as serum bilirubin, serum glutamic-oxaloacetic transaminase (SGOT), and serum glutamate pyruvate transaminase (SGPT) ≤ 2 times the upper limit of normal (ULN), and creatinine ≤ 1.5 times the ULN.
9. Patient must have an ECOG score of ≤ 2.
10. The patient has a negative human immunodeficiency virus antibody (HIV) test result.

Exclusion Criteria:

A patient will be ineligible for study participation if any of the following criteria are met:

1. The patient has a history of an allergic reaction or significant sensitivity to Panhematin®.
2. The patient has taken or used any investigational drug or device in the 30 days prior to screening.
3. The patient has chronic myelomonocytic leukemia (CMML).
4. The patient has a history of deep vein thrombosis or known hypercoagulable state.
5. The patient has a history of a pre-existing medical condition that, in the opinion of the investigator, will interfere with the participation in the study.
6. The patient has poor peripheral venous access, if central venous access is not available.
7. The patient has an uncontrolled active infection.
8. The patient has positive test results for hepatitis B surface antigen, and hepatitis C virus antibody.
9. The patient has any other condition or prior therapy that, in the opinion of the Investigator, would make the patient unsuitable for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2007-05; Primary Completion 2008-12 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jamile Shammo, MD, Principal Investigator — Rush University Medical Center
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States

REFERENCES:
- [Background] Aul C, Germing U, Gattermann N, Minning H. Increasing incidence of myelodysplastic syndromes: real or fictitious? Leuk Res. 1998 Jan;22(1):93-100. doi: 10.1016/s0145-2126(97)00089-1. PMID 9585086
- [Background] Aul C, Giagounidis A, Germing U. Epidemiological features of myelodysplastic syndromes: results from regional cancer surveys and hospital-based statistics. Int J Hematol. 2001 Jun;73(4):405-410. doi: 10.1007/BF02994001. PMID 11503953
- [Background] Catenacci DV, Schiller GJ. Myelodysplasic syndromes: a comprehensive review. Blood Rev. 2005 Nov;19(6):301-19. doi: 10.1016/j.blre.2005.01.004. PMID 15885860
- [Background] Cheson BD, Bennett JM, Kantarjian H, Pinto A, Schiffer CA, Nimer SD, Lowenberg B, Beran M, de Witte TM, Stone RM, Mittelman M, Sanz GF, Wijermans PW, Gore S, Greenberg PL; World Health Organization(WHO) international working group. Report of an international working group to standardize response criteria for myelodysplastic syndromes. Blood. 2000 Dec 1;96(12):3671-4. PMID 11090046
- [Background] Dhar GJ, Bossenmaier I, Cardinal R, Petryka ZJ, Watson CJ. Transitory renal failure following rapid administration of a relatively large amount of hematin in a patient with acute intermittent porphyria in clinical remission. Acta Med Scand. 1978;203(5):437-43. doi: 10.1111/j.0954-6820.1978.tb14903.x. PMID 665312
- [Background] Fibach E, Kollia P, Schechter AN, Noguchi CT, Rodgers GP. Hemin-induced acceleration of hemoglobin production in immature cultured erythroid cells: preferential enhancement of fetal hemoglobin. Blood. 1995 May 15;85(10):2967-74. PMID 7537986
- [Background] Greenberg P, Cox C, LeBeau MM, Fenaux P, Morel P, Sanz G, Sanz M, Vallespi T, Hamblin T, Oscier D, Ohyashiki K, Toyama K, Aul C, Mufti G, Bennett J. International scoring system for evaluating prognosis in myelodysplastic syndromes. Blood. 1997 Mar 15;89(6):2079-88. PMID 9058730
- [Background] Mauritzson N, Albin M, Rylander L, Billstrom R, Ahlgren T, Mikoczy Z, Bjork J, Stromberg U, Nilsson PG, Mitelman F, Hagmar L, Johansson B. Pooled analysis of clinical and cytogenetic features in treatment-related and de novo adult acute myeloid leukemia and myelodysplastic syndromes based on a consecutive series of 761 patients analyzed 1976-1993 and on 5098 unselected cases reported in the literature 1974-2001. Leukemia. 2002 Dec;16(12):2366-78. doi: 10.1038/sj.leu.2402713. PMID 12454741
- [Background] McHale CM, Winter PC, Lappin TR. Erythroid gene expression is differentially regulated by erythropoietin, haemin and delta-aminolaevulinic acid in UT-7 cells. Br J Haematol. 1999 Mar;104(4):829-37. doi: 10.1046/j.1365-2141.1999.01269.x. PMID 10192446
- [Background] Monette FC, Holden SA. Hemin enhances the in vitro growth of primitive erythroid progenitor cells. Blood. 1982 Aug;60(2):527-30. PMID 7093531
- [Background] Panhematin® Product Prescribing Information. Abbott Laboratories, August 2000 Edition
- [Background] Porter PN, Meints RH, Mesner K. Enhancement of erythroid colony growth in culture by hemin. Exp Hematol. 1979 Jan;7(1):11-6. PMID 428474
- [Background] Rund D, Ben-Yehuda D. Therapy-related leukemia and myelodysplasia: evolving concepts of pathogenesis and treatment. Hematology. 2004 Jun;9(3):179-87. doi: 10.1080/10245330410001701503. PMID 15204099
- [Background] Thompson JE, Luger SM. The role of hematopoietic stem cell transplantation in myelodysplastic syndrome. Oncology (Williston Park). 2005 Apr;19(4):533-42; discussion 542-4, 547-8. PMID 15934520
- [Background] Timonen TT, Kauma H. Therapeutic effect of heme arginate in myelodysplastic syndromes. Eur J Haematol. 1992 Nov;49(5):234-8. doi: 10.1111/j.1600-0609.1992.tb00054.x. PMID 1473585
- [Background] Volin L, Ruutu T, Knuutila S, Tenhunen R. Heme arginate treatment for myelodysplastic syndromes. Leuk Res. 1988;12(5):423-31. doi: 10.1016/0145-2126(88)90062-8. PMID 3379975
- [Background] Williamson PJ, Kruger AR, Reynolds PJ, Hamblin TJ, Oscier DG. Establishing the incidence of myelodysplastic syndrome. Br J Haematol. 1994 Aug;87(4):743-5. doi: 10.1111/j.1365-2141.1994.tb06733.x. PMID 7986716
- [Background] Vidaza® Product Prescribing Information. Pharmion Corporation, 5-18-04 Edition

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between 5/2007 and 10/2008, 6 patients were enrolled on trial and were treated at Rush university medical center.
Groups:
- Group 1: Panhematin treatment arm
Period: Overall Study
Arm/Group | Group 1
Started | 6
Completed | 5
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Group 1
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 5
Age, Continuous [Mean (Full Range); unit: years] | 73 (0) [64 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 5
Region of Enrollment [Number; unit: participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: Safety and Tolerability of Panhematin®.
Description: Number of patients with no adverse events.
Time Frame: participants were followed during therapy with panhematin, and up to six months post completion of therapy, average of 8 months.
Measure: Number; unit: participants
Arm/Group | Group 1
Number analyzed (Participants) | 6
participants | 6

2. Secondary Outcome: Number of Patients Demonstrating Hematological Improvement to Panhematin® at Week 4.
Description: Hematological improvement (HI)
  Major:
  HI-Erythroid:>2 g/dL rise in hemoglobin, or transfusion independence HI-Neutrophil: Absolute increase of >500/mm3, or >100% increase HI-Platelet: Absolute increase of >30,000, or transfusion independence
  Minor:
  HI-Erythroid:1 to 2 g/dL increase in hemoglobin or 50% decrease in transfusion dependence.
  HI-P: For patients with pretreatment platelet count < 100,000/mm3, ≥ 50% increase with a net increase > 10,000/mm3 but < 30,000/mm3.
  HI-N: For patients with pretreatment ANC < 1500/mm3, ≥ 100% increase, but < 500/mm3 increase.
Time Frame: 4 weeks after initiation of treatment with Panhematin
Measure: Number; unit: participants
Arm/Group | Group 1
Number analyzed (Participants) | 5
participants | 0

3. Primary Outcome: Response Rate ( CR+PR) at Week 8, Based on the IWG Criteria for Response Assessment ( 2000 Version)
Description: Complete response(CR): <5% blasts in the bone marrow,with normal maturation of all cell lines, Hemoglobin >11 g/dL, neutrophils>1500/mm3 platelets>100,000/mm3.
  Partial response (PR): >50% decrease in blasts, or less advanced IPSS than pretreatment value, same hematological parameters as in CR.
  Stable disease (SD): No evidence of disease progression in bone marrow, stable peripheral blood counts failure: Increase in bone marrow blast percentage, progression to more advanced IPSS than pretreatment and worsening of cytopenias.
  (Cheson, 2000)
Time Frame: After 8 weeks of therapy with panhematin
Measure: Number; unit: Participants
Arm/Group | Group 1
Number analyzed (Participants) | 5
Participants | 0

4. Secondary Outcome: Hematological Improvement Rate at Week 8 as Defined by the IWG 2000 Criteria for Response Assessment, 2000 Version
Time Frame: At 8 weeks from start of therapy
Measure: Number; unit: participants
Arm/Group | Group 1
Number analyzed (Participants) | 5
participants | 1

ADVERSE EVENTS:
Time Frame: All adverse events occuring from the time of subject signing informed consent through 30 days post completion of study were collected. about 8 months period.
Arm/Group | Group 1
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No